CLINICAL TRIAL: NCT00675779
Title: Comparison of Pain Relief and Inflammatory Status in Women With Surgically Confirmed Endometriosis Treated With Atorvastatin, Oral Contraceptive or Combined Oral Contraceptives and Atorvastatin: Open Randomized Controlled Trial
Brief Title: Efficacy Study of Atorvastatin in Pelvic Pain Relief in Women With Endometriosis
Acronym: EndoStatin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: University of California, Davis (Other); Biomet Polska Sp. z.o.o. (Industry)
Responsible Party: Robert Z. Spaczynski, MD PhD, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204-08
Record Dates: First submitted 2008-05-05; First posted 2008-05-12 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Endometriosis; Pain
Keywords: endometriosis; atorvastatin; oral; contraception; pain; relief; pelvic pain in women with endometriosis
MeSH Terms: conditions — Endometriosis; Pain | interventions — Contraceptives, Oral; ethinyl estradiol-desogestrel combination; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): oral contraceptive + atorvastatin
  Interventions: Drug: atorvastatin + oral contraceptive
- 1 (Active Comparator): oral contraceptive
  Interventions: Drug: oral contraceptive (Mercilon)

INTERVENTIONS:
Drug: oral contraceptive (Mercilon) — oral contraceptive (20ug EE, 150ug DSG) 1 tablet a day p.o. for 21 days with 7 day break for 6 months
  Other Names: Mercilon (Organon Schering-Plough, Poland)
  Arms: 1
Drug: atorvastatin + oral contraceptive — atorvastatin 20mg po a day for 6 months + oral contraceptive (20ug EE, 150ug DSG) 1 tablet po a day for 21 days with 7 day break for 6 months
  Other Names: Atrox 20 (Biofarm sp. z o.o. , Poznan, Poland)
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether atorvastatin (alone or in combination with oral contraceptive) is effective in treatment of pelvic pain and inflammatory response in women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent
* premenopausal women aged 18-45
* clinical signs and symptoms of endometriosis for minimum 3 months with endometriosis confirmed at laparoscopy or laparotomy within last 4 months - 5 years (preferably with histological confirmation)
* pain symptoms of moderate intensity (dysmenorrhoea + dyspareunia + nonmenstrual pelvic pain > 6 points on Biberoglu & Behrman scale [1981])
* no clinical signs of sexually transmitted disease

Exclusion Criteria:

* cancer of the ovary, adrenals, endometrium, uterine cervix, breasts
* pregnancy or lactation
* unexplained uterine/cervical bleeding
* hormonal therapy within last 3 months (for GnRH analogs 6 months)
* irregular menses (> 35 days) or secondary amenorrhoea (>3 months)
* other chronic disease affecting pelvic or abdominal cavity (including PID, ulcerating colitis , Crohn's disease, recurrent interstitial cystitis)
* sexually transmitted disease (gonorrhoea, Chlamydia)
* uncontrolled diabetes mellitus type I or II, VTE or other contraindications to medicine used in the study
* chronic therapy with CYP3A4 inhibitors (including ketoconazole, erythromycin and others)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-11 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
pain relief | 3,6,12 months

SECONDARY OUTCOMES:
inflammatory status | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoni J Duleba, MD, Study Chair — University of California, Davies, USA; Leszek Pawelczyk, MD PhD, Study Director — Poznan University of Medical Sciences, Poland
Locations (1):
- Poznan University of Medical Sciences, Department of Gynecology and Obstetrics, Poznan, Poland